CLINICAL TRIAL: NCT02878707
Title: The Neuroprotective Effects of Dexmedetomidine During Brain Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201605056MIFA
Record Dates: First submitted 2016-08-15; First posted 2016-08-25 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2016-08

CONDITIONS: Brain Tumor; Cerebrovascular Disorders
MeSH Terms: conditions — Brain Neoplasms; Cerebrovascular Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX (Experimental): Intraoperative intravenous infusion of dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): Intraoperative intravenous infusion of 0.9% saline
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Intraoperative dexmedetomidine infusion

SUMMARY:
Dexmedetomidine (DEX) is a Alpha-2 specific agonist, is a common ICU sedation medication. In brain tumor resection craniotomy, it is proven to be effective in improving postoperative hypertension and tachycardia, mitigates postoperative nausea and vomiting and relives postoperative pain. In addition, many animal experiments show that DEX inhibits the proapoptosis in the mitochondrial in vivo and therefore avoids neuronal injury. It is also reported to be neuroprotective to isoflurane-induced neurotoxicity and to improve cerebral focal ischemic region (penumbra). However, the neuroprotective effects were never investigated clinically in patients undergoing brain tumor resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective craniotomy for supratentorial brain tumor resection or cerebral vascular surgery
* age between 20 to 80 yr

Exclusion Criteria:

* Fever, elevated white blood cell or C-reactive protein
* Impaired liver function, eg. AST or ALT >100; liver cirrhosis > Child B class
* Impaired renal function, cGFR< 60 ml/min/1.73 m2
* Cardiac dysfunction, such as heart failure > NYHA class II

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative neurological complications | during postoperative period of hospital admission, approximately 10 days by estimation

SECONDARY OUTCOMES:
Number of participants with postoperative delirium | during postoperative period of hospital admission, approximately 10 days by estimation
Serum biomarkers changes | Between preoperative baseline and postoperative day one.
  biomarkers related to neuroinflammation and neuronal injury, such as HMGB1 and GFAP
Intraoperative haemodynamic profile | during intraoperative perioid, approximately 4-6 hours by estimation

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, MD, Principal Investigator — Anesthesiology Department, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen PH, Tsuang FY, Lee CT, Yeh YC, Cheng HL, Lee TS, Chang YW, Cheng YJ, Wu CY. Neuroprotective effects of intraoperative dexmedetomidine versus saline infusion combined with goal-directed haemodynamic therapy for patients undergoing cranial surgery: A randomised controlled trial. Eur J Anaesthesiol. 2021 Dec 1;38(12):1262-1271. doi: 10.1097/EJA.0000000000001532. PMID 34101714